CLINICAL TRIAL: NCT03065140
Title: Muscle Fat Compartments and Turnover as Determinant of Insulin Sensitivity - the MISTY Study
Brief Title: Muscle Fat Compartments and Turnover as Determinant of Insulin Sensitivity
Acronym: MISTY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16/NS/0024
Record Dates: First submitted 2016-12-07; First posted 2017-02-27 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): Healthy volunteers will undergo the following:
  * CPEX with/without stable isotope infusion
  * Muscle biopsies
  * Magnetic Resonance Spectroscopy Followed by a period of detraining.
  They will then undergo the following:
  * CPEX with/without stable isotope infusion
  * Muscle biopsies
  * Magnetic Resonance Spectroscopy
  Interventions: Other: Training or detraining
- Diabetic Patients (Experimental): Diabetic patients will undergo the following:
  * CPEX with/without stable isotope infusion
  * Muscle biopsies
  * Magnetic Resonance Spectroscopy They will then undergo a supervised training period.
  They will then undergo the following:
  * CPEX with/without stable isotope infusion
  * Muscle biopsies
  * Magnetic Resonance Spectroscopy
  Interventions: Other: Training or detraining

INTERVENTIONS:
Other: Training or detraining — A period of detraining or a supervised exercise program.
  Other Names: Detraining or training

SUMMARY:
Early research found that high levels of fat within muscle meant poorer control of blood sugar. However, more recent research has shown that athletes have similar levels of fat within muscle, but in contrast, they have very good control of blood sugar. The investigators are not sure why this is and want to find out if the fat within muscle can be changed to improve blood sugar control, as good blood sugar control reduces the risk of heart disease, diabetes and stroke.

DETAILED DESCRIPTION:
Higher levels of triglycerides (TG) and diacylglycerols (DAG) are found in skeletal muscle of patients with obesity/diabetes as well as in trained athletes. Despite similar metabolic storage, patients and athletes have opposite insulin sensitivity phenotypes and an explanation for this is lacking. The investigators' objective is to understand how these fat compartments can be beneficially modulated to improve insulin resistance and cardio-metabolic risk. The investigators will investigate if either structural differences (saturated versus unsaturated balance of TG and DAG side-chains) or different handling abilities (fast versus slow lipid pool turnover) will be induced by exercise capacity interventions in athletes and in diabetic patients. In a longitudinal study pre- and post-exercise, the investigators will use novel, non-invasive 1H-Magnetic Resonance Spectroscopy to benchmark the saturated/unsaturated compartments against skeletal muscle biopsies for the first time and stable isotope analysis for fat compartments' rate of turnover.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients, aged between 20-65, diagnosed as per WHO criteria, diet controlled or diet and any of the following oral hypoglycemics: metformin, sulphonylureas, glitazones, gliptins, acarbose, but not requiring insulin for controlling of blood glucose.
* Trained, athletic healthy controls, aged 18 and over.
* Participant who is willing and able to give informed consent for participation in the study.
* Able to perform exercise testing.

Exclusion Criteria:

* Any history of known coronary artery disease.
* Other endocrine conditions
* Impaired renal function defined as eGFR<60mls/min/1.73m2
* Known resting/24 hour BP >160/100mmHg
* Participants on ACE inhibitors
* Participants on PPAR agonists
* Participants on omega 3 fatty acids
* The existence of any medical or surgical condition that in the judgement of the investigators may interfere with the exercise regime, FA metabolism or may compromise the safety of the subject
* Presence of other significant concomitant heart diseases such as ischaemic, valvular, pericardial heart disease or cardiomyopathy, skeletal muscle disorders
* Healthy volunteers that are on any chronic medication that in the judgment of the investigators is likely to affect the outcome of the study
* Significant asthma
* Significant pulmonary disease
* Participants unable to cycle on the ergometer
* Unable to perform exercise testing (e.g. prosthetic limbs)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Non-invasive 1H Magnetic Resonance Spectroscopy of vastus lateralis | One Hour
  Assessment of energetics of vastus lateralis by MRS

SECONDARY OUTCOMES:
Saturated and unsaturated lipid pool turnover examined by stable isotopes | One hour
  Lipid pool turnover as examined by stable isotope infusion

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, MD, Principal Investigator — University of Aberdeen Employee
Locations (1):
- Cardiac Research Office, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobley GE, Holtrop G, Bremner DM, Calder AG, Milne E, Johnstone AM. Impact of short term consumption of diets high in either non-starch polysaccharides or resistant starch in comparison with moderate weight loss on indices of insulin sensitivity in subjects with metabolic syndrome. Nutrients. 2013 Jun 10;5(6):2144-72. doi: 10.3390/nu5062144. PMID 23752495
- [Background] Wilson FA, van den Borne JJ, Calder AG, O'Kennedy N, Holtrop G, Rees WD, Lobley GE. Tissue methionine cycle activity and homocysteine metabolism in female rats: impact of dietary methionine and folate plus choline. Am J Physiol Endocrinol Metab. 2009 Apr;296(4):E702-13. doi: 10.1152/ajpendo.90670.2008. Epub 2009 Jan 13. PMID 19141688
- [Background] Phillips DI, Caddy S, Ilic V, Fielding BA, Frayn KN, Borthwick AC, Taylor R. Intramuscular triglyceride and muscle insulin sensitivity: evidence for a relationship in nondiabetic subjects. Metabolism. 1996 Aug;45(8):947-50. doi: 10.1016/s0026-0495(96)90260-7. PMID 8769349
- [Background] Kumashiro N, Erion DM, Zhang D, Kahn M, Beddow SA, Chu X, Still CD, Gerhard GS, Han X, Dziura J, Petersen KF, Samuel VT, Shulman GI. Cellular mechanism of insulin resistance in nonalcoholic fatty liver disease. Proc Natl Acad Sci U S A. 2011 Sep 27;108(39):16381-5. doi: 10.1073/pnas.1113359108. Epub 2011 Sep 19. PMID 21930939
- [Background] Goodpaster BH, He J, Watkins S, Kelley DE. Skeletal muscle lipid content and insulin resistance: evidence for a paradox in endurance-trained athletes. J Clin Endocrinol Metab. 2001 Dec;86(12):5755-61. doi: 10.1210/jcem.86.12.8075. PMID 11739435
- [Background] Amati F, Dube JJ, Alvarez-Carnero E, Edreira MM, Chomentowski P, Coen PM, Switzer GE, Bickel PE, Stefanovic-Racic M, Toledo FG, Goodpaster BH. Skeletal muscle triglycerides, diacylglycerols, and ceramides in insulin resistance: another paradox in endurance-trained athletes? Diabetes. 2011 Oct;60(10):2588-97. doi: 10.2337/db10-1221. Epub 2011 Aug 26. PMID 21873552
- [Background] Manco M, Mingrone G, Greco AV, Capristo E, Gniuli D, De Gaetano A, Gasbarrini G. Insulin resistance directly correlates with increased saturated fatty acids in skeletal muscle triglycerides. Metabolism. 2000 Feb;49(2):220-4. doi: 10.1016/s0026-0495(00)91377-5. PMID 10690948
- [Background] Anastasiou CA, Kavouras SA, Lentzas Y, Gova A, Sidossis LS, Melidonis A. Diabetes mellitus is associated with increased intramyocellular triglyceride, but not diglyceride, content in obese humans. Metabolism. 2009 Nov;58(11):1636-42. doi: 10.1016/j.metabol.2009.05.019. Epub 2009 Jul 16. PMID 19615699
- [Background] Coen PM, Dube JJ, Amati F, Stefanovic-Racic M, Ferrell RE, Toledo FG, Goodpaster BH. Insulin resistance is associated with higher intramyocellular triglycerides in type I but not type II myocytes concomitant with higher ceramide content. Diabetes. 2010 Jan;59(1):80-8. doi: 10.2337/db09-0988. Epub 2009 Oct 15. PMID 19833891
- [Background] Bergman BC, Perreault L, Hunerdosse DM, Koehler MC, Samek AM, Eckel RH. Increased intramuscular lipid synthesis and low saturation relate to insulin sensitivity in endurance-trained athletes. J Appl Physiol (1985). 2010 May;108(5):1134-41. doi: 10.1152/japplphysiol.00684.2009. Epub 2010 Mar 18. PMID 20299618
- [Background] King DS, Dalsky GP, Clutter WE, Young DA, Staten MA, Cryer PE, Holloszy JO. Effects of exercise and lack of exercise on insulin sensitivity and responsiveness. J Appl Physiol (1985). 1988 May;64(5):1942-6. doi: 10.1152/jappl.1988.64.5.1942. PMID 3292505
- [Background] Dube JJ, Amati F, Toledo FG, Stefanovic-Racic M, Rossi A, Coen P, Goodpaster BH. Effects of weight loss and exercise on insulin resistance, and intramyocellular triacylglycerol, diacylglycerol and ceramide. Diabetologia. 2011 May;54(5):1147-56. doi: 10.1007/s00125-011-2065-0. Epub 2011 Feb 17. PMID 21327867
- [Background] Dube JJ, Amati F, Stefanovic-Racic M, Toledo FG, Sauers SE, Goodpaster BH. Exercise-induced alterations in intramyocellular lipids and insulin resistance: the athlete's paradox revisited. Am J Physiol Endocrinol Metab. 2008 May;294(5):E882-8. doi: 10.1152/ajpendo.00769.2007. Epub 2008 Mar 4. PMID 18319352
- [Background] Goodpaster BH, Katsiaras A, Kelley DE. Enhanced fat oxidation through physical activity is associated with improvements in insulin sensitivity in obesity. Diabetes. 2003 Sep;52(9):2191-7. doi: 10.2337/diabetes.52.9.2191. PMID 12941756
- [Background] Summers SA, Nelson DH. A role for sphingolipids in producing the common features of type 2 diabetes, metabolic syndrome X, and Cushing's syndrome. Diabetes. 2005 Mar;54(3):591-602. doi: 10.2337/diabetes.54.3.591. PMID 15734832
- [Background] Bruce CR, Thrush AB, Mertz VA, Bezaire V, Chabowski A, Heigenhauser GJ, Dyck DJ. Endurance training in obese humans improves glucose tolerance and mitochondrial fatty acid oxidation and alters muscle lipid content. Am J Physiol Endocrinol Metab. 2006 Jul;291(1):E99-E107. doi: 10.1152/ajpendo.00587.2005. Epub 2006 Feb 7. PMID 16464906
- [Background] Brechtel K, Niess AM, Machann J, Rett K, Schick F, Claussen CD, Dickhuth HH, Haering HU, Jacob S. Utilisation of intramyocellular lipids (IMCLs) during exercise as assessed by proton magnetic resonance spectroscopy (1H-MRS). Horm Metab Res. 2001 Feb;33(2):63-6. doi: 10.1055/s-2001-12407. PMID 11294494
- [Background] Boden G, Lebed B, Schatz M, Homko C, Lemieux S. Effects of acute changes of plasma free fatty acids on intramyocellular fat content and insulin resistance in healthy subjects. Diabetes. 2001 Jul;50(7):1612-7. doi: 10.2337/diabetes.50.7.1612. PMID 11423483
- [Background] Machann J, Etzel M, Thamer C, Haring HU, Claussen CD, Fritsche A, Schick F. Morning to evening changes of intramyocellular lipid content in dependence on nutrition and physical activity during one single day: a volume selective 1H-MRS study. MAGMA. 2011 Feb;24(1):29-33. doi: 10.1007/s10334-010-0233-8. Epub 2011 Jan 7. PMID 21213017
- [Background] Kelley DE, Goodpaster B, Wing RR, Simoneau JA. Skeletal muscle fatty acid metabolism in association with insulin resistance, obesity, and weight loss. Am J Physiol. 1999 Dec;277(6):E1130-41. doi: 10.1152/ajpendo.1999.277.6.E1130. PMID 10600804
- [Background] Perreault L, Bergman BC, Hunerdosse DM, Playdon MC, Eckel RH. Inflexibility in intramuscular triglyceride fractional synthesis distinguishes prediabetes from obesity in humans. Obesity (Silver Spring). 2010 Aug;18(8):1524-31. doi: 10.1038/oby.2009.454. Epub 2009 Dec 24. PMID 20035285
- [Background] Lizcano JM, Alessi DR. The insulin signalling pathway. Curr Biol. 2002 Apr 2;12(7):R236-8. doi: 10.1016/s0960-9822(02)00777-7. No abstract available. PMID 11937037
- [Background] Delibegovic M, Bence KK, Mody N, Hong EG, Ko HJ, Kim JK, Kahn BB, Neel BG. Improved glucose homeostasis in mice with muscle-specific deletion of protein-tyrosine phosphatase 1B. Mol Cell Biol. 2007 Nov;27(21):7727-34. doi: 10.1128/MCB.00959-07. Epub 2007 Aug 27. PMID 17724080
- [Background] Bence KK, Delibegovic M, Xue B, Gorgun CZ, Hotamisligil GS, Neel BG, Kahn BB. Neuronal PTP1B regulates body weight, adiposity and leptin action. Nat Med. 2006 Aug;12(8):917-24. doi: 10.1038/nm1435. Epub 2006 Jul 16. PMID 16845389
- [Background] Boesch C, Machann J, Vermathen P, Schick F. Role of proton MR for the study of muscle lipid metabolism. NMR Biomed. 2006 Nov;19(7):968-88. doi: 10.1002/nbm.1096. PMID 17075965
- [Background] Hock A, Fuchs A, Boesiger P, Kollias SS, Henning A. Electrocardiogram-triggered, higher order, projection-based B(0) shimming allows for fast and reproducible shim convergence in spinal cord (1)H MRS. NMR Biomed. 2013 Mar;26(3):329-35. doi: 10.1002/nbm.2852. Epub 2012 Oct 13. PMID 23065738
- [Background] Hock A, MacMillan EL, Fuchs A, Kreis R, Boesiger P, Kollias SS, Henning A. Non-water-suppressed proton MR spectroscopy improves spectral quality in the human spinal cord. Magn Reson Med. 2013 May;69(5):1253-60. doi: 10.1002/mrm.24387. Epub 2012 Jun 28. PMID 22745036
- [Background] Kuhlmann J, Neumann-Haefelin C, Belz U, Kalisch J, Juretschke HP, Stein M, Kleinschmidt E, Kramer W, Herling AW. Intramyocellular lipid and insulin resistance: a longitudinal in vivo 1H-spectroscopic study in Zucker diabetic fatty rats. Diabetes. 2003 Jan;52(1):138-44. doi: 10.2337/diabetes.52.1.138. PMID 12502504
- [Background] Ye Q, Danzer CF, Fuchs A, Wolfrum C, Rudin M. Hepatic lipid composition differs between ob/ob and ob/+ control mice as determined by using in vivo localized proton magnetic resonance spectroscopy. MAGMA. 2012 Oct;25(5):381-9. doi: 10.1007/s10334-012-0310-2. Epub 2012 Mar 23. PMID 22441585
- [Background] van Loon LJ, Koopman R, Manders R, van der Weegen W, van Kranenburg GP, Keizer HA. Intramyocellular lipid content in type 2 diabetes patients compared with overweight sedentary men and highly trained endurance athletes. Am J Physiol Endocrinol Metab. 2004 Sep;287(3):E558-65. doi: 10.1152/ajpendo.00464.2003. Epub 2004 May 27. PMID 15165998
- [Background] Liu Y, Li J, Zhang Z, Tang Y, Chen Z, Wang Z. Effects of exercise intervention on vascular endothelium functions of patients with impaired glucose tolerance during prediabetes mellitus. Exp Ther Med. 2013 Jun;5(6):1559-1565. doi: 10.3892/etm.2013.1064. Epub 2013 Apr 11. PMID 23837031
- [Background] Dudzinska W, Lubkowska A, Jakubowska K, Suska M, Skotnicka E. Insulin resistance induced by maximal exercise correlates with a post-exercise increase in uridine concentration in the blood of healthy young men. Physiol Res. 2013;62(2):163-70. doi: 10.33549/physiolres.932355. Epub 2012 Dec 13. PMID 23234409
- [Background] Alibegovic AC, Sonne MP, Hojbjerre L, Bork-Jensen J, Jacobsen S, Nilsson E, Faerch K, Hiscock N, Mortensen B, Friedrichsen M, Stallknecht B, Dela F, Vaag A. Insulin resistance induced by physical inactivity is associated with multiple transcriptional changes in skeletal muscle in young men. Am J Physiol Endocrinol Metab. 2010 Nov;299(5):E752-63. doi: 10.1152/ajpendo.00590.2009. Epub 2010 Aug 24. PMID 20739510
- [Background] Ducommun S, Wang HY, Sakamoto K, MacKintosh C, Chen S. Thr649Ala-AS160 knock-in mutation does not impair contraction/AICAR-induced glucose transport in mouse muscle. Am J Physiol Endocrinol Metab. 2012 May 15;302(9):E1036-43. doi: 10.1152/ajpendo.00379.2011. Epub 2012 Feb 7. PMID 22318952
- [Background] ECG-Triggered and Respiratory Gated Image Based B0 Shimming for Single Voxel Spectroscopy of the Myocardium at 3T. 21st Annual Meeting and Exhibition of the International Society for Magnetic Resonance in Medicine (ISMRM 2013), Salt Lake City, UT, USA. 2013